CLINICAL TRIAL: NCT00744822
Title: Vibration Response Imaging (VRI) in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Deep Breeze (Industry)
Responsible Party: Merav Gat, Director of Clinical Affairs, Deep Breeze Ltd.
Other Study IDs: 4066
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Last update posted 2008-09-01 (Estimated); Status verified 2005-12

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Infections; Graft Rejection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a prospective, multi-center study. 50 lung transplant recipients will be enrolled in the study. Subjects will be selected from lung transplant recipients, who have undergone single or double lung transplantation during the last six months These patients will undergo a baseline VRI recording prior to the interventional procedure and a follow-up VRI at 1 hour after the interventional procedure. Furthermore, the patients will be recorded at the designated follow-up periods of 1, 3 and 6-month (+ 7 days) post-baseline visit, as well as before and 1 hour after any recurrent interventional procedure

DETAILED DESCRIPTION:
* Study participants will be patients who have undergone lung transplantation during the last 6 months and are in a stable clinical position at the time of enrollment.
* Patients who meet the study inclusion and exclusion criteria will be enrolled in the study.
* The enrolled patients will be recorded with the VRI at each occurrence in which the standard procedures are performed:

  * Baseline after study enrollment (VRI Recording 1 + standard evaluations).
  * At each follow-up visit [1, 3, 6 months after baseline visit] during the 6 month follow-up period of the study (VRI Recordings + standard evaluations (if possible)).
  * In the event of bronchoscopic intervention, then before the interventional procedure (VRI Recording 1 + standard evaluations) and before any recurrent interventional procedures (VRI Recordings + standard evaluations) during the course of the study (6-month follow-up period).
  * 1 hour after all bronchoscopic interventional procedures.
  * In the event of an unanticipated visit, then a VRI recording will be performed (VRI Recordings + standard evaluations).
* All subjects will be recorded according to a standard procedure; moreover, it is essential that for each subject repeatable recordings will be performed in the same manner (i.e. breathing manner and matrix placement). Each VRI recording session will take ~15 minutes [the actual recording is ~2 minutes for placement and breathing/recording].
* Standard evaluation procedures may include any of the following:

  * Lung function tests (this test is required at all visits)
  * Physical examination
  * Bronchoscopy (e.g. transbronchial biopsy)
  * CT-imaging
  * Chest x-ray
  * V/Q Scan (Baseline visit for single lung transplantation)
  * Blood gases (this test is required at all visits)
  * Blood tests

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be entered into the study:

1. Able and willing to read, understand, and provide written Informed Consent
2. Male or Female in the age range of 18-65 years
3. Subject is a lung transplant recipient who underwent single or double lung transplantation within the last 6 months
4. BMI > 19
5. Height of >1.55 meters
6. Stable clinical condition at study baseline evaluation

Exclusion Criteria:

Any of the following will exclude the subject from study:

1. Intubated patients
2. Chest wall deformation
3. Spine deformation (including severe scoliosis)
4. Hirsutism
5. Potentially contagious skin lesion on the back
6. Skin lesion that would interfere with sensor placement
7. Cardiac pacemaker or implantable defibrillator
8. Patient is pregnant as confirmed with urine pregnancy test
9. Colonization of multi-resistant bacteria (MRSA) If the subject meets all of the inclusion criteria and none of the exclusion criteria, he/she is eligible to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 lung transplant recipients will be enrolled in the study. Subjects will be selected from lung transplant recipients, who have undergone single or double lung transplantation during the last six months
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to evaluate the ability of VRI lung images in single lung or double lung transplant recipients to assist the physician in detecting risk factors associated with lung transplantation during the six-month follow-up period | 6 months

SECONDARY OUTCOMES:
The secondary objective is to compare evaluations of the lung VRI images with the results of other evaluation techniques [i.e. PFT, chest X-ray]. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany